CLINICAL TRIAL: NCT06364826
Title: Gemcitabine, Sintilimab, Bevacizumab Plus IMRT in Patients With Cisplatin Ineligible Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Sintilimab Combination Therapy Plus IMRT in Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaozhong, chief physicians, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-202403
Record Dates: First submitted 2024-03-26; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: locoregionally advanced Nasopharyngeal carcinoma; sintilimab; bevacizumab; IMRT
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — sintilimab; Bevacizumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sintilimab, bevacizumab, gemcitabine (Experimental): Patients will receive induction therapy (sintilimab + bevacizumab + gemcitabine, Q3W, 3 cycles) followed by IMRT+ Sintilimab. Consolidation therapy with sintilimab continued after radiotherapy until disease progression, intolerable toxicity, death, or the subject's decision to withdraw from the study, with a total treatment period of no more than 12 cycles.
  Interventions: Drug: Sintilimab, bevacizumab, gemcitabine; Radiation: IMRT

INTERVENTIONS:
Drug: Sintilimab, bevacizumab, gemcitabine — This is a prospective, single-center, single-arm, phase II clinical study. The study was intended to include patients with locoregionally advanced nasopharyngeal cancer identified by histology or cytology, who signed informed consent and met the screening criteria to enter the study. Patients will receive induction therapy (sintilimab + bevacizumab + gemcitabine, Q3W, 3 cycles) followed by IMRT+ Sintilimab. Consolidation therapy with sintilimab continued after radiotherapy until disease progression, intolerable toxicity, death, or the subject's decision to withdraw from the study, with a total treatment period of no more than 12 cycles.
Radiation: IMRT — IMRT

SUMMARY:
This is a prospective, single-center, single-arm, phase II clinical study. The study was intended to include patients with locoregionally advanced nasopharyngeal cancer identified by histology or cytology, who signed informed consent and met the screening criteria to enter the study. Patients will receive induction therapy (sintilimab + bevacizumab + gemcitabine, Q3W, 3 cycles) followed by IMRT+ Sintilimab. Consolidation therapy with sintilimab continued after radiotherapy until disease progression, intolerable toxicity, death, or the subject's decision to withdraw from the study, with a total treatment period of no more than 12 cycles.

DETAILED DESCRIPTION:
Platinum deplatinization has been extensively explored in patients with posterior nasopharyngeal carcinoma who have received multiple platinum treatments, including target-free combination, GEP, etc. Our center also published in 2022 CSCO a study on the preliminary efficacy of pembrolizumab combined with gemcitabine in the first-line treatment of metastatic NPC with or without cisplatin or anlotinib. Enrolled patients were treated with pembrolizumab + anlotinib +GP (group A), pembrolizumab +GP (group B), and pembrolizumab + anlotinib +G (group C), with ORR of 80% (4/5), 80% (4/5), and 100% (7/7), respectively. Among them, there were 1 CR and 6 PR in group C. Compared to group B, group C with anlotinib in place of cisplatin showed a better safety profile with fewer grade 3 adverse reactions (57.1% vs 100%). In summary, we designed this study to evaluate the efficacy and safety of gemcitabine, sintilimab and bevacizumab combined with IMRT in patients with advanced nasopharyngeal carcinoma not suitable for platinum-based treatment, and to explore new therapeutic approaches for patients with advanced stage nasopharyngeal carcinoma who cannot tolerate platinum therapy or are unwilling to receive platinum therapy.

This is a prospective, single-center, single-arm, phase II clinical study. The study was intended to include patients with locoregionally advanced nasopharyngeal cancer identified by histology or cytology, who signed informed consent and met the screening criteria to enter the study. Patients will receive induction therapy (sintilimab + bevacizumab + gemcitabine, Q3W, 3 cycles) followed by IMRT+ Sintilimab. Consolidation therapy with sintilimab continued after radiotherapy until disease progression, intolerable toxicity, death, or the subject's decision to withdraw from the study, with a total treatment period of no more than 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign a written informed consent before implementing any procedures related to the trial; 2. No gender limitation, age ≥18 years old, ≤75 years old; 3. Histological or cytological determination of advanced nasopharyngeal carcinoma assessed by the investigator without any treatment (stage III-IVA, except T3N0M0); 4. Not suitable for platinum therapy (patients > 70 years old, PS > 2, hearing impairment, renal insufficiency (creatinine clearance < 50ml/min) or grade 1 neuropathy;2023 CSCO Guidelines for the Diagnosis and Treatment of Head and Neck Tumors) or patients do not receive platinum therapy; 5. The ECOG PS score is 0-1; 6. According to the solid tumor efficacy evaluation criteria (RECIST version 1.1), there is at least one radiographically measurable lesion; 7. Expected survival time > 6 months; 8. Adequate organ function.

Exclusion Criteria:

* 1. Patients with uncured malignancies other than advanced nasopharyngeal carcinoma diagnosed within 5 years prior to initial administration (excluding radical basal cell carcinoma of the skin, squamous epithelial carcinoma of the skin, and/or carcinoma in situ after radical resection); 2. Is currently participating in an interventional clinical study, or has received other investigational drugs or used investigational devices within 4 weeks prior to initial dosing; 3. Previous treatment with anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs that target another stimulus or synergistically inhibit T cell receptors (e.g., CTLA-4, OX-40, CD137); 4. Previously received anti-angiogenic therapy, including but not limited to anti-angiogenic monoclonal antibodies, anti-angiogenic TKI, etc.; 5. Received systemic systemic treatment with proprietary Chinese medicines with anti-tumor indications or immunomodulatory drugs (including thymosin, interferon, interleukin) within 2 weeks before the first administration; 6. An active autoimmune disease requiring systemic treatment (e.g. with disease-modifying drugs, glucocorticoids, or immunosuppressants) has occurred within 2 years prior to first administration.Replacement therapies (such as thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy; 7. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation; 8. Known active ingredients or excipients of Sintilimab and bevacizumab in this study, and allergic patients to chemotherapy drugs in this study; 9. Has not fully recovered from toxicity and/or complications caused by any intervention before starting treatment (i.e., ≤ grade 1 or baseline, excluding weakness or hair loss); 10. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive); 11. Other researchers did not consider it appropriate to study enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-22 (Estimated); Primary Completion 2026-04-22 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
3-year Event-free survival rate | 3 years
  The time between the start of treatment and the first occurrence of any of the following events: disease progression, local or distant recurrence, death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Objective Response Rate | 3 years
  Proportion of total subjects in complete response (CR) and partial response (PR)
Disease Control Rate | 3 years
  Proportion of subjects defined as complete response (CR), partial response (PR), and stable disease (SD)
Progression-Free Survival | 3 years
  The time between the start of treatment and first radiographic disease progression or death, whichever occurs first
Overall survival | 3 years
  The time of treatment until the subject dies from any cause
adverse events(AEs) | 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

OTHER OUTCOMES:
biomarkers | 3 years
  To evaluate the relationship between biomarkers and response

IPD SHARING:
Plan to Share IPD: No